CLINICAL TRIAL: NCT05349006
Title: A Randomized, Placebo-controlled Phase 3 Trial of Azathioprine for the Prevention of Relapse in Myelin-oligodendrocyte-glycoprotein (MOG)-Antibody Associated Disease
Brief Title: Azathioprine in MOGAD
Acronym: MOGwAI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL21_1065
Record Dates: First submitted 2022-04-15; First posted 2022-04-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Central Nervous System Inflammation; MOG-IgG Associated Disease
Keywords: MOGAD; azathioprine; optic neuritis; myelitis; neuromyelitis optica; MOG-IgG associated disease
MeSH Terms: conditions — Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Optic Neuritis; Myelitis; Neuromyelitis Optica | interventions — Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azathioprine (Experimental): Azathioprine, dose related to weight (100 mg for weight ≤ 50 kg and 150 mg for weight > 50 kg), oral, daily
  Associated to oral corticosteroid, prednisone : 40 mg per day during three months, and progressively tapered during three months until stop (- 30 mg during 15 days, 20mg during 15 days, 15 mg during 15 days, 10 mg during 15 days, 5 mg during 15 days and introduction of hydrocortisone 20 mg + Stop prednisone; hydrocortisone 20mg during 15 days, Stop hydrocortisone)
  Interventions: Drug: Azathioprine
- Placebo (Placebo Comparator): Placebo, once a day, oral, number of caps related to weight
  Associated to oral corticosteroid: prednisone 40 mg per day during three months and progressively tapered during three months until stop (- 30 mg during 15 days, 20mg during 15 days, 15 mg during 15 days, 10 mg during 15 days, 5 mg during 15 days and introduction of hydrocortisone 20 mg + Stop prednisone; hydrocortisone 20mg during 15 days, Stop hydrocortisone)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azathioprine — Dose related to weigh (100 mg for weight ≤ 50 kg and 150 mg for weight > 50 kg) = 2 to 4 50mg oral caps, daily, during all the study period
  Arms: Azathioprine
Other: Placebo — Dose related to weigh (100 mg for weight ≤ 50 kg and 150 mg for weight > 50 kg) = 2 to 4 50mg oral caps, daily, during all the study period
  Arms: Placebo

SUMMARY:
MOG-IgG associated disease (MOGAD) is a rare inflammatory disease of the central nervous system recently described. Initially reported as monophasic, data from incident cohorts suggests that around 50% of adult patients with MOG-Ab may relapse within the first two years of the disease, with most of relapses occurring early after disease onset.

No randomized controlled trial has ever been performed and therapeutic guidelines for this disease remain unclear especially after a single event. In short-sized and mainly retrospective study, azathioprine, an immunosuppressant drug, have showed promising results on preventing the risk of relapse in MOGAD patients.

The hypothesis is that the initiation of a treatment after a first attack of MOGAD should prevent further relapse and disability accrual. The investigators propose herein the first randomized controlled trial in MOGAD, to evaluate the efficacy of azathioprine to prevent relapses, after a first attack, in a placebo double-blinded design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First attack of documented acute demyelinating syndrome of the central nervous system, within the past 3 months, whatever the severity or the clinical phenotype
* Tested positive for MOG-Ab, confirmed in a centralized lab (Lyon referral centre)
* Ability of the subject to understand the purpose and risks of the study and provide signed and dated written informed consent.
* Patients should be beneficiary of health care coverage under the social security system
* Female patients of childbearing potential should have effective contraception throughout the course of treatment and for at least three months after stopping treatment.

Exclusion Criteria:

* Hypersensitivity to azathioprine or steroids
* Active infections or cancer (including tuberculosis, hepatitis, herpes and VZV)
* Psychosis not controlled by treatment
* Seriously impaired bone marrow functions: Lymphocyte count < 1000/ml and or Polynuclear neutrophil count < 1500/ml
* Seriously impaired hepatic functions: ALT and/or AST > 3N
* Seriously impaired renal functions: GFR < 29 ml/min/1.73m²
* Any live vaccine in the past 3 months or planned during the RCT and RCT+6months
* Thiopurine methyltransferase (TPMT) phenotype deficient or intermediate, with enzymatic activity < 16 nmol/h/ml
* Unable to complete an MRI (e.g. due to pacemaker, severe claustrophobia, hypersensitivity to contrast media, or who lack adequate peripheral venous access)
* Necessary use of a xanthine oxidase inhibitor (Allopurinol, Oxipurinol, Thiopurinol, Febuxotat,…)
* Necessary use of angiotensin-converting-enzyme inhibitor, cotrimoxazole, cimetidine and indometacine
* Necessary use of an aminosalicylate derivates
* Necessary use of any another immunosuppressive therapy, different than azathioprine, or steroids
* Necessary use of cytotoxic therapy
* Necessary use of any other medical illness or disability that, in the opinion of the investigator, would compromise effective trial participation
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy is use within 5 half-lives prior to baseline. Participation in a non- interventional study can be allowed as long as this participation does not interfere with this protocol or is not likely to affect the subject's ability to comply with the protocol.
* For subjects coming back from strongyloidiasis endemic regions, a parasitology screening examination will be performed on faeces, and that appropriate treatment will be performed prior to administration of corticosteroids
* Patients with Lesch Nyhan syndrome
* Asian patients (probable mutation of the gene NUDT1)
* Female subjects who have a positive a positive urinary or blood pregnancy test result, are pregnant or are currently breast feeding
* Inability to comply with study requirements
* Person under legal protection or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2029-12-12 (Estimated)

PRIMARY OUTCOMES:
Time to first relapse (in days), comparing azathioprine-treated vs placebo-treated patients during a randomized control period of a maximum of three years. | During a randomized control period of a maximum of three years
  A definite relapse will be defined as such:
  * When a patient is diagnosed as experiencing a relapse by the local investigator, the anonymized file will be reviewed within 4 days by a second investigator neurologist, not aware of the randomization group nor of the center treating the patient.
  * If this second neurologist also considers the patient as experiencing a relapse, the patient will be considered as relapsing for the main analysis.
  * If the second neurologist disagrees, the opinion of a third neurologist will be asked and the majority opinion will be retained.
  As to ensure a maximum of homogeneity, we also propose a protocol-defined criteria for a MOGAD relapse, validated by the steering committee and available to every investigator (see Annex 2).

SECONDARY OUTCOMES:
Number and type of adverse events, including serious adverse events, related to azathioprine and/or steroids and placebo | : During a randomized control period of a maximum of three years
Evaluation of global disability at 36 months | at baseline and at 36 months
  Global disability at 36 months assessed by EDSS: The EDSS scale is a method of quantifying disability and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of patients with inflammatory disorders of the central nervous system. The EDSS scale ranges from 0 to 10 in 0.5-unit increments (20 values) that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Evaluation of global disability at 36 months | at baseline and at 36 months
  Worsening from baseline to 36 months of the EDSS
Evaluation of global disability at 36 months | at baseline and at 36 months
  Ambulation status at 36 months assessed by the Ambulation Score. Scoring is based on a measurement of the distance the patient is able to walk (in meters) and then classified in 12 levels.
Evaluation of global disability at 36 months | at baseline and at 36 months
  Worsening from baseline to 36 months of the Ambulation Score.
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Best-corrected high contrast visual acuity at 36 months measured (each eye tested separately) using the standard Snellen chart or equivalent.
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Worsening from baseline to 36 months of visual disability assessed by change of the best- corrected high-contrast visual acuity using the standard Snellen chart or equivalent (each eye tested separately).
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Best-corrected low-contrast visual acuity at 36 months using the Sloan Charts at 2.5%, in each eye.
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Worsening from baseline to 36 months of low-contrast visual acuity using the Sloan Charts at 2.5%, in each eye.
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Inner retinal layers thicknesses at 36 months assessed by the spectral domain OCT (each eye tested separately)
Evaluation of visual disability at 36 months | at baseline and at 36 months
  Worsening from baseline to 36 months of the peripapillary retinal nerve fiber layer thickness (μm) and the ganglion cell complex thickness (μm) assessed with spectral domain OCT (each eye tested separately).
Quality of life will be assessed using the EuroQOL EQ-5D-3L at 36 months | at 36 months
  https://euroqol.org
Compliance to treatment | During a randomized control period of a maximum of three years
  percentage of untaken pills (left in the blisters) regarding each patient
Exploratory radiological features | at baseline and at 36 months
  Description, and comparison between the two groups, of worsening of MRI (brain and spinal cord and visual) from baseline to 36 months assessed by number of new/enlarging T2 lesions
Exploratory radiological features | at baseline and at 36 months
  Description and comparison between the two groups of worsening of MRI (brain and/or spinal cord and/or visual) from baseline to 36 months assessed by number of new T1 gadolinium enhancing lesions
Exploratory biological features | at screening, at 6 months, at 12 months, at 36 months and in case of a relapse
  In each group of treatment, association between MOG-Ab titer at first episode and the risk of relapse
Exploratory biological features | at screening, at 6 months, at 12 months, at 36 months and in case of a relapse
  In each group of treatment, association between MOG-Ab titer at onset and the level of global disability assessed by the EDSS at 36 months.
Exploratory biological features | at screening, at 6 months, at 12 months, at 36 months and in case of a relapse
  In each group of treatment, prognostic value of longitudinal MOG-Ab-titers to predict relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Romain MARIGNIER, MD PhD, Study Director — Hospices Civils de Lyon
Locations (17):
- France (17):
  - Department of Neurology, CHU de Bordeaux - GH Pellegrin, Bordeaux
  - Department of Neurology, CHU of Lille, Hospital Roger Salengro, Lille
  - Department of Neuro Ophthalmology, CHU of Lyon, Neurology Hospital Pierre Wertheimer, Lyon
  - Service de Neurologie sclérose en plaques, pathologies de la myéline et neuro-inflammation - Centre de référence des maladies inflammatoires rares du cerveau et de la moelle (MIRCEM) - Hôpital Neurologique Pierre Wertheimer - Hospices Civils de Lyon, Lyon
  - Department of Neurology University hospital Timone, Marseille
  - Department of Neurology Montpellier Universitary Hospital, Montpellier
  - CHRU de Nancy Hôpital Central, Nancy
  - Department of Neurology, Hôpital Pasteur 2, Nice
  - Department of Neurology, Hôpital Caremeau, Nîmes
  - National Hospital of Vision (15-20), Paris
  - Department of Neurology APHP, Pitié Salpêtrière Hospital, Paris
  - Department of Neurology. Hôpital A. Fondation Rothschild, Paris
  - Department of Neurology, CHU de Rennes, Rennes
  - Department of Neurology, CHU de Rouen, Rouen
  - Department of Neurology, Hôpital g. Et r. Laennec, Saint-Herblain
  - Department of Neurology, Hôpital Hautepierre, Strasbourg
  - Department of Neurology, Toulouse Universitary Hospital, Toulouse